CLINICAL TRIAL: NCT04762069
Title: A Multicenter, Open-Label Study With a Randomized Control Arm of the Efficacy, Safety, and Pharmacokinetics of Intravenously Infused Berubicin in Adult Patients With Recurrent Glioblastoma Multiforme After Failure of Standard First Line Therapy
Brief Title: A Study of Berubicin in Adult Subjects With Recurrent Glioblastoma Multiforme
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CNS Pharmaceuticals, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNS-201
Record Dates: First submitted 2020-11-11; First posted 2021-02-21 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma Multiforme, Adult
Keywords: Glioblastoma Multiforme; Glioblastoma; Brain Cancer; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Lomustine

STUDY DESIGN:
Intervention Model Description: Open-Label Study with a Randomized Control Arm
Who Masked: Outcomes Assessor
Masking Description: Response and progression outcomes are evaluated by a blinded central reviewer for each patient according to RANO criteria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Berubicin (Experimental): Berubicin intravenously infused will be administered at a dose of 7.1 mg/m2 as free base as a 2 hour intravenous (IV) infusion once daily for 3 consecutive days followed by 18 days off study drug (each cycle = 21 days)
  Each treatment cycle is 21 days. Subjects will be allowed to continue on treatment at the discretion of the Investigator if there is no evidence of disease progression and the subject is not experiencing unacceptable toxicity as well as if both the subject and Investigator agree that further therapy is in the subject's best interest.
  Interventions: Drug: Berubicin
- Lomustine (CCNU, CeeNU®, or Gleostine®) capsules (Active Comparator): Lomustine (CCNU, CeeNU®, or Gleostine®) capsules will be administered at the institutionally-approved dose and regimen or per the full prescribing information/summary of product characteristics.
  Interventions: Drug: Lomustine

INTERVENTIONS:
Drug: Berubicin — Berubicin HCl is a novel synthetic anthracycline with a chemical structure similar to doxorubicin HCl, a cytotoxic anthracycline topoisomerase II inhibitor isolated from cultures of Streptomyces peucetius var. caesius.
  Other Names: Berubicin Hydrochloride
  Arms: Berubicin
Drug: Lomustine — Lomustine is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug. This medication is classified as an "alkylating agent.
  Other Names: Lomustine Capsules; CCNU; CeeNU; Gleostine
  Arms: Lomustine (CCNU, CeeNU®, or Gleostine®) capsules

SUMMARY:
This is an open-label, multicenter, randomized, parallel, 2-arm, efficacy and safety study. Patients with GBM after failure of standard first line therapy will be randomized in a 2:1 ratio to receive berubicin or lomustine for the evaluation of OS. Additional endpoints will include response and progression outcomes evaluated by a blinded central reviewer for each patient according to RANO criteria.

A pre-planned, non-binding futility analysis will be performed after approximately 30 to 50% of all planned patients have completed the primary endpoint at 6 months. This review will include additional evaluation of safety as well as secondary efficacy endpoints. Enrollment will not be paused during this interim analysis.

DETAILED DESCRIPTION:
Berubicin is one of the first anthracyclines that crosses the blood brain barrier and overcomes drug resistance (i.e. it is not a substrate for multi-drug resistant/breast cancer resistant transporters). A Phase 1 clinical trial of berubicin in patients with primary CNS malignancies demonstrated a durable response (one subject alive 13+ years) as well as stable disease in heavily pretreated patients. Therefore, this phase 2 study is designed to further evaluate Berubicin's activity in patients with rGBM after treatment with standard of care.

ELIGIBILITY:
Patients will be eligible for the study if they meet all of the following inclusion criteria and none of the exclusion criteria.

Inclusion criteria

1. Written informed consent from the patient or their legally authorized representative (LAR) prior to any study-related procedure, and willing and able to comply with the protocol and aware of the investigational nature of this study.
2. At least 18 years of age.
3. KPS score of ≥ 60
4. A confirmed GBM diagnosis must be based on local review of tumor tissue from the initial biopsy, surgery, or re-resection. A formal pathology report confirming GBM is acceptable. It is not a requirement for slides to be sent to a central reviewer.
5. Recurrent or progressive GBM as evaluated by central review applying RANO criteria on contrast MRI scans of the Baseline/Screening MRI scan obtained up to six weeks prior to C1D1 and a historical scan taken before the Baseline/Screening scan that meets at least 1 of the following criteria:

   1. In the case of measurable disease, progression will be documented by ≥ 25% increase in the sum of the perpendicular diameter products (SPDPs) of the measurable contrast-enhancing (target) lesions or any new measurable lesions.
   2. If the SPDPs cannot be reliably estimated due to the lesion's complex conspicuity, shape, and contrast enhancement pattern, the volume of all measurable and non-measurable lesions may be used instead, applying the same threshold (≥ 25% increase) to confirm disease progression.
   3. In the case of non-measurable lesions in the historical scan, any transformation into measurable lesions (≥10 mm in both maximum perpendicular diameters) in the Baseline/Screening scan will be evidence of progression.
   4. If there are only non-measurable (non-target) lesions in the Baseline/Screening scan, additional lesions/sites will be considered evidence of progression based on the historical scan. Patients with new cerebrospinal fluid (CSF) seeding will not be considered eligible.
   5. If historical scans are unavailable, a radiology report of a scan taken before the Baseline/Screening scan documenting the SPDPs from a previous scan of the enhancing disease or its volume can be used by the central reviewer to assess eligibility if it demonstrates the quality standards and acquisition guidelines required.
   6. If the scan obtained during standard of care (prior to initiation of formal clinical screening and patient enrollment) is being used as the Baseline/Screening scan and does not entirely conform to central reader quality standards and acquisition guidelines (ie, artifacts or missing sequences), this can be used for the purpose of inclusion if the central reader in discussion with the sponsor and PI agree it provides evidence based on standard clinical practices of recurrence or progression.
   7. Patients at first progression who are treated by re-resection or biopsy to confirm progression do not require measurable disease at their post-operative screening scan as their Baseline/Screening scan. These patients must be medically stable after the procedure as assessed by the PI and have the Baseline/Screening scan available by 7 days before starting treatment.
6. The tumor is localized supratentorially with no leptomeningeal (local or distant), spinal or CSF metastases, and no ventricular invasion (explicit documentation of the disease progression that would be problematic in evaluating the efficacy of this drug).
7. O[6] methylguanine-DNA methyltransferase (MGMT) methylation status must be available; results of routinely used methods for MGMT methylation testing (eg, methylation-specific polymerase chain reaction or quantitative polymerase chain reaction) are acceptable.
8. No more than 1 prior line of treatment (eg, surgery followed by radiation with concomitant chemotherapy, followed by adjuvant chemotherapy is considered as 1 line of treatment). In addition, treatment with tumor treating fields (TTFields; Optune) is acceptable if provided as first line therapy prior to progression or recurrence of disease.
9. A second debulking surgery, additional radiation or gamma knife surgery during the first line treatment or after progression, and for which the investigator does not suspect pseudoprogression is acceptable, as long as no chemotherapy or immunotherapy has been provided.
10. Recovery from toxicity/side effects of all prior therapy to Grade 1 or less, subject to the investigator's discretion, except for alopecia; the following time intervals from previous treatments are required to be eligible:

    1. 12 weeks from the completion of radiation (to reduce risk of pseudoprogression), unless progression is confirmed by biopsy
    2. 4 weeks from the end of any previous of chemotherapy
    3. 2 weeks from tumor biopsy if wound completely healed
    4. 4 weeks from any major surgery (maximal debulking surgery, either gross total resection or partial resection), gamma knife surgery or significant traumatic injury. Any surgery incisions or wounds must be completely healed
11. A stable or decreasing dose of corticosteroids (or none) for brain edema for at least 5 days prior to baseline MRI and enrollment in the study to document disease progression such that changes in the MRI are not related to the use of corticosteroids.
12. Eligible for chemotherapy based on adequate bone marrow function and organ function within 2 weeks of study treatment as defined by the following laboratory guidelines, subject to the investigator's discretion:

    1. Hematopoietic function: total white blood cell (WBC) count ≥3 × 103/µL, absolute neutrophil count (ANC) ≥1.5 × 10³/µL, platelet count ≥75 × 10³/µL, hemoglobin ≥10 g/dL
    2. Hepatic function: bilirubin ≤1.5 × × the upper limit of normal (ULN) (excluding Gilberts Syndrome, for which bilirubin must be ≤4 × ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 × ULN, and alkaline phosphatase ≤2.5 × ULN
    3. Renal function: serum creatinine ≤1.5 × ULN or for patients with creatinine levels above the ULN, estimated creatinine clearance of ≥60 mL/min, calculated using the Cockcroft-Gault equation35
    4. Activated partial thromboplastin time (aPTT) ≤1.5 × ULN
13. Women of childbearing potential must agree to practice a highly effective method of contraception beginning at least 28 days before the start of treatment until at least 6.25 months after the last dose of study drug. Male study patients and their female sexual partners of childbearing potential must agree to practice a highly effective method of contraception starting from the time of informed consent until at least 3.5 months (no less than 104 days) after the last dose of study drug.

    1. A woman of childbearing potential is defined as a woman who is not permanently sterilized or postmenopausal. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.
    2. Women of childbearing potential must have a negative serum or urine pregnancy test at Screening.
    3. A highly effective method of birth control is defined as one which results in a low failure rate (ie, less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. For patients using a hormonal contraceptive method, information regarding all medications being administered to the patient and their potential effects on the contraceptive should be addressed.
14. Patients with prior malignancies must be disease-free for ≥5 years. Curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; or prostate cancer as well as benign tumors that will not interfere with the treatment plan at the time of screening are allowed.

Exclusion Criteria

1. Unable or not willing to comply with the protocol regulations.
2. Any additional chemotherapy (including but not limited to TMZ or immunotherapy) for recurrent or progressive GBM after a first line treatment.
3. Prior treatment with bevacizumab.
4. Prior treatment with lomustine.
5. Known to have an IDH mutation prior to enrollment
6. Screening/Baseline MRI showing a mass effect defined as significant compression of the ventricular system and/or a midline shift with associated clinical symptoms deemed inappropriate for the patient to enter a clinical trial. If there is otherwise asymptomatic compression and/or midline shift and the patient fulfills all other criteria, these patients are considered eligible.
7. Any condition (medical, social, psychological) that would prevent adequate information and follow-up, including but not limited to clinically relevant psychiatric disorders, legal incapacity, dementia, adults protected by law or altered mental status.
8. Presence of poorly controlled seizures, defined as occurring despite SOC or requiring hospitalization.
9. Prior anthracycline cumulative dose more than 550 mg/m2.
10. Heart disease:

    1. LVEF <50%
    2. Unstable angina
    3. CHF with New York Heart Association (NYHA) classification of 3 or 4
    4. Patients with baseline QT/QTc interval >480 msec, a history of additional risk factors for torsades de pointes (TdP) (eg, heart failure, hypokalemia, family history of long QT syndrome) and using concomitant medications that significantly prolong the QT/QTc interval
    5. History of myocardial infarction within 12 months of enrollment
    6. Severe arrhythmia not controlled by medication
11. Uncontrolled hypertension (systolic blood pressure [BP] >150 mmHg and/or diastolic BP >100 mmHg) sustained over 2 measurements.
12. Known to be positive for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV), human immunodeficiency virus (HIV), COVID-19 (currently positive at time of screening), or any other acute viral, bacterial, or fungal infection (testing not required unless symptomatic or suspected disease).
13. Patients with any other uncontrolled intercurrent medical conditions, including but not limited to diabetes mellitus or chronic obstructive pulmonary disease that have not been well controlled by medical management over the prior 3 months are ineligible unless approved by the sponsor.
14. Women who are lactating or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Through study completion an average of 4 years.
  To assess the effect of berubicin compared with lomustine on overall survival (OS) in adult patients with GBM that has recurred or progressed after standard initial therapy

SECONDARY OUTCOMES:
Progression Free Survival | Through study completion an average of 4 years.
  To assess the effect of berubicin on progression free survival per Response Assessment in Neuro-Oncology (RANO) criteria in patients with GBM after failure of standard first line therapy
Event Free Survival | Through study completion an average of 4 years.
  To assess the effect of berubicin on event free survival (EFS) defined as the length of time from the initiation of study drug administration to disease progression, death, or discontinuation of treatment for any reason (eg, toxicity, intolerance, disease-related conditions, or failure to respond)
Overall Response Rate | Through study completion an average of 4 years.
  To assess the effect of berubicin on overall response rates (ORR) in adult patients with GBM after failure of standard first line therapy
Safety of the Recommended Phase 2 Dose of Berubicin | From signing of informed consent until until 28 days after the last dose of berubicin and 42 days after the last dose of lomustine, or until the patient receives any additional therapy for their disease (whichever comes first).
  To assess the safety of the recommended Phase 2 dose of berubicin by the incidence and severity of adverse events (AEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 5.0.
Plasma Pharmacokinetics Cmax | Through study completion an average of 4 years.
  Maximum plasma concentration of Berubicin
Plasma Pharmacokinetics tmax | Through study completion an average of 4 years.
  Time from each dose to reach the maximum plasma concentration
Plasma Pharmacokinetics AUC0-tau | Through study completion an average of 4 years.
  Area under the plasma concentration-time curve from time 0 to Tau, where Tau is the dosing interval, calculated by the linear up/ linear down trapezoidal method
Plasma Pharmacokinetics AUC0-last | Through study completion an average of 4 years.
  Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration calculated by the linear up/log linear down trapezoidal method
Plasma Pharmacokinetics AUC0-∞ | Through study completion an average of 4 years.
  Area under the plasma concentration-time curve from time 0 to infinite time, calculated as the sum of AUC0-last and Clast/λz, where Clast is the last observed quantifiable concentration
Plasma Pharmacokinetics t1/2 | Through study completion an average of 4 years.
  elimination half-life associated with the terminal slope (λz) of the log-linear drug concentration-time curve, calculated as ln(2)/λz
Plasma Pharmacokinetics CL | Through study completion an average of 4 years.
  apparent total body clearance
Plasma Pharmacokinetics Vz | Through study completion an average of 4 years.
  apparent volume of distribution
Plasma Pharmacokinetics Css | Through study completion an average of 4 years.
  Average concentration, calculated as the geometric mean of concentrations over the 72-hour dosing interval
Plasma Pharmacokinetics Rac | Through study completion an average of 4 years.
  The accumulation ratio calculated as AUC0-tau (3rd dose) / AUC0-tau (1st dose)

OTHER OUTCOMES:
Karnofsky Performance Status | Through study completion an average of 4 years.
  Evaluate changes in Karnofsky Performance Status (KPS) score between arms
Evaluate changes in patient-reported outcomes | Through study completion an average of 4 years.
  Evaluate changes in patient-reported outcomes between arms.
Explore the effect of O[6] methylguanine-DNA methyltransferase (MGMT) methylation | Through study completion an average of 4 years.
  explore the effect of O[6] methylguanine-DNA methyltransferase (MGMT) methylation status on response to berubicin and comparison of theses subsets between arms
Impact of re-resection | Through study completion an average of 4 years.
  Impact of re-resection on outcomes
Use of bevacizumab | Through study completion an average of 4 years.
  Use of bevacizumab between the arms.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Silberman, MD, PhD, Study Chair — CNS Pharmaceuticals, Inc.
Locations (48):
- United States (32):
  - University of Arkansas, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Los Angeles, California
  - University of California Irvine, Orange, California
  - University of Califonia San Diego Moores Cancer Center, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Saint John's Cancer Institute at Providence Saint John's Health Center, Santa Monica, California
  - HCA Healthcare Research Institute, Englewood, Colorado
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Baptist Miami, Miami, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Rush University Cancer Center, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Tulane Cancer Center Clinic, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - UMass (ACC) - Hollings Cancer Center (HCC), Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Rutgers University, Piscataway, New Jersey
  - Atlantic Healthcare, Summit, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Providence Health, Portland, Oregon
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Texas Oncology PA, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Huntsman Cancer Center, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- France (7):
  - Hopital Pierre Wertheimer, Lyon
  - Hopital de La Timone, Marseille
  - Institut de Recherche en Cancerologie de Montpellier, Montpellier
  - Hopital Pitie-Salpetriere, Paris
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
  - nstitut Universitaire du Cancer de Toulouse-, Toulouse
  - Institut de Cancerologie Gustave-Roussy, Villejuif
- Italy (2):
  - Servizio Sanitario Regionale Emilia-Romagna - Azienda USL di Bologna - Ospedale Bellaria, Bologna
  - Istituto Clinico Humanitas, Milan
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga Carlos Haya, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Study data will be shared with WPD Pharmaceuticals, Inc., sub-licensee of Berubicin.